CLINICAL TRIAL: NCT03626896
Title: A FIH Feasibility Study to Evaluate the Safety of Transient Disruption of Blood-brain Barrier in Recurrent Glioblastoma Multiforme (GBM) Patients Using NaviFUS System
Brief Title: Safety of BBB Disruption Using NaviFUS System in Recurrent Glioblastoma Multiforme (GBM) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NaviFUS Corporation (Industry)
Collaborators: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: NF-2017-01
Record Dates: First submitted 2018-08-07; First posted 2018-08-13 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2018-08

CONDITIONS: Glioblastoma Multiforme; Brain Tumor; Glioblastoma; Glioma; Neoplasms; Neoplasms, Nerve Tissue
Keywords: BBB disruption; NaviFUS System; Focused Ultrasound; GBM
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms; Glioma; Neoplasms; Neoplasms, Nerve Tissue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NaviFUS System (Experimental): NaviFUS System: dose escalation focus ultrasound to transiently disrupt BBB
  Interventions: Device: NaviFUS System

INTERVENTIONS:
Device: NaviFUS System — BBB Disruption by FUS in recurrent GBM Other Name: Neuronavigation-guided focus ultrasound system

SUMMARY:
This study is to evaluate the safety and find the tolerated ultrasound dose of transient opening of the blood-brain barrier (BBB) by using the NaviFUS System in recurrent GBM patients.

DETAILED DESCRIPTION:
This is a feasibility, open-label, single-arm, and dose escalation study. Eligible patients will be enrolled through the process of informed consent. Patients will be assigned into different dose groups generated from the NaviFUS System to transiently open the BBB in patients with recurrent GBM who will undergo surgery within 2 weeks. The focused ultrasound (FUS) dose is selected based on the results of pre-clinical Good Laboratory Practice (GLP) safety studies as well as other non-GLP primate studies. This study will evaluate the safety and the tolerated ultrasound dose of temporary disruption of the BBB in patients with recurrent GBM. To find the tolerated ultrasound dose, the data and safety monitoring board (DSMB) will review the study data and provide the recommendations regarding continuation, termination, or other modifications of the study based on evaluation of observed adverse effects of the intervention. The extent and magnitude of BBB opening will be evaluated using of dynamic contrast-enhanced MRI (DCE-MRI).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with recurrent GBM and will undergo surgery
* Able to give written informed consent for the participation in the trial
* Adult male/female patients > 20 years of age
* Patients if already on radiotherapy, a gap of 7 days shall be maintained between the last day of radiotherapy and the day of screening
* Patients if already on the steroids treatment, then should be on a stable dose of steroids for at least 7 days prior to screening
* Body mass index (BMI) ≥17 kg / m2
* Patients with life expectancy ≥ 3 months
* Able to comply with study requirements in the opinion of the investigator
* Adequate hepatic, renal, coagulation, and hematopoietic function

  * Hemoglobin ≥ 10 g/dL
  * Platelets ≥ 100,000/mm3
  * Neutrophils ≥ 1,500/mm3
  * Normal creatinine clearance ≥ 50mL/min
  * Alanine transaminase (ALT) < 3 x upper limit of normal (ULN)
  * Aspartate transaminase (AST) < 3 x ULN
  * Prothrombin time ≤ 1.2 x ULN
  * International Normalized Ratio (INR) < 1.5
  * Bilirubin < 2 x ULN
* Patients with the ROI for FUS exposure are located close to the cortex with at least 20 mm distance beneath the skull bone and the ROI is not in the deep center brain with crucial brain functions, such as in the region of brain stem, or motor or speech regions
* The Karnofsky performance status (KPS) in the patient must be > 60

Exclusion Criteria:

* Patients at screening visit have arteriovenous malformation (AVM) or cerebral aneurysm
* Use of any recreational drugs or history of drug addiction
* Pregnant or breast-feeding women
* The receipt of an investigational drug, or participation in a drug research study within a period of one month prior to the first FUS exposure
* Known sensitivity/allergy to MRI contrast agents, CT contrast agents, SonoVue®, or any of its components
* Any other condition that, in the investigator's judgment, might increase the risk to the patients or decrease the chance of obtaining satisfactory data needed to achieve the objectives of the study
* Abnormal baseline findings considered by the investigator to indicate conditions that might affect study endpoints
* Patients who have hemorrhage or cyst within the ROI
* Severe hypertension at screening (diastolic blood pressure > 100 mmHg on medication)
* Receiving anticoagulant (e.g. warfarin) or antiplatelet (e.g. aspirin) therapy within one week prior to study treatment or drugs known to increase risk or hemorrhage (e.g. Avastin) within one month prior to study treatment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-08-17 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2019-06-19 (Actual)

PRIMARY OUTCOMES:
Number and severity of AE | 45 days
  Safety of transient opening of the BBB by using the NaviFUS System

SECONDARY OUTCOMES:
Tolerated dose of FUS with the NaviFUS System for transient disruption of the BBB | 7 days post-FUS
  Dose escalation study using FUS
Quantify the BBB disruption following BBB disruption by the NaviFUS System | 1 day
  Dynamic T1 contrast-enhanced MRI

CONTACTS AND LOCATIONS:
Overall Officials: Kuo-Chen Wei, M.D., Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Linkou Chang Gung Memorial Hospital, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Background] Wei KC, Tsai HC, Lu YJ, Yang HW, Hua MY, Wu MF, Chen PY, Huang CY, Yen TC, Liu HL. Neuronavigation-guided focused ultrasound-induced blood-brain barrier opening: a preliminary study in swine. AJNR Am J Neuroradiol. 2013 Jan;34(1):115-20. doi: 10.3174/ajnr.A3150. Epub 2012 Jun 21. PMID 22723060
- [Background] McDannold N, Zhang Y, Vykhodtseva N. Blood-brain barrier disruption and vascular damage induced by ultrasound bursts combined with microbubbles can be influenced by choice of anesthesia protocol. Ultrasound Med Biol. 2011 Aug;37(8):1259-70. doi: 10.1016/j.ultrasmedbio.2011.04.019. Epub 2011 Jun 8. PMID 21645965
- [Background] Liu HL, Wai YY, Chen WS, Chen JC, Hsu PH, Wu XY, Huang WC, Yen TC, Wang JJ. Hemorrhage detection during focused-ultrasound induced blood-brain-barrier opening by using susceptibility-weighted magnetic resonance imaging. Ultrasound Med Biol. 2008 Apr;34(4):598-606. doi: 10.1016/j.ultrasmedbio.2008.01.011. Epub 2008 Mar 3. PMID 18313204
- [Background] Hynynen K, McDannold N, Sheikov NA, Jolesz FA, Vykhodtseva N. Local and reversible blood-brain barrier disruption by noninvasive focused ultrasound at frequencies suitable for trans-skull sonications. Neuroimage. 2005 Jan 1;24(1):12-20. doi: 10.1016/j.neuroimage.2004.06.046. PMID 15588592
- [Background] Wei KC, Chu PC, Wang HY, Huang CY, Chen PY, Tsai HC, Lu YJ, Lee PY, Tseng IC, Feng LY, Hsu PW, Yen TC, Liu HL. Focused ultrasound-induced blood-brain barrier opening to enhance temozolomide delivery for glioblastoma treatment: a preclinical study. PLoS One. 2013;8(3):e58995. doi: 10.1371/journal.pone.0058995. Epub 2013 Mar 19. PMID 23527068